CLINICAL TRIAL: NCT06894095
Title: Dongzong Cardiovascular Bio-imaging Registry Study
Acronym: DAILY
Status: Recruiting | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhang longjiang,MD, Principal Investigator (PI): Zhang Longjiang; Co-PI: Tang Chunxiang, Jinling Hospital, China
Other Study IDs: 2023NZKY-018-02
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases; Multi-omics; Living Environments; Pulmonary-cardiovascular Imaging
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 10 ml of blood and 2 ml of saliva will be collected from each patient for the evaluation of conventional laboratory parameters. A portion of the sample will be analyzed for established clinical biomarkers, including lipid profiles, blood biochemistry, inflammatory markers, liver function, and renal function, among others. Additionally, the residual biological specimens will be employed for sequencing in various omics fields, including genomics, transcriptomics, proteomics, metabolomics, microbiomics, and other omics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The DAILY project is a large-scale, multicenter, prospective initiative designed to establish a comprehensive bio-imaging database that integrates multidimensional data, including living environments, psychosocial and cognitive assessments, advanced lung and cardiovascular imaging, multi-omics profiles, clinical medication and surgical records, and health outcomes. Leveraging this extensive, multiscale dataset, the project aims to elucidate the intricate interplay between genetic biology and environmental factors in driving downstream biological alterations, thereby shaping lung and cardiovascular structural and functional phenotypes, and ultimately influencing the onset and progression of cardiovascular diseases (CVD). Through a systematic exploration and understanding of this complex network, the project seeks to identify critical intervention points and develop innovative strategies for the prevention and management of CVD.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) are the leading cause of global mortality, representing a major public health challenge that threatens life and health both presently and in the foreseeable future. The reduction of modifiable risk factors remains a powerful and essential strategy, however, the application of clinical risk scores has demonstrated limited efficacy in significantly reducing cardiovascular events. In recent years, the emergence of multi-omics has provided novel insights into the prevention and management of CVD, offering opportunities to deeply understand its drivers at the genetic and biological levels. Nevertheless, the clinical utility and widespread adoption of these approaches face significant challenges, primarily due to two critical factors: First, multi-omics datasets, particularly GWAS datasets, exhibit a pronounced Eurocentric bias; second, the vast array of multi-omics indicators cannot be effectively integrated with living environments and diseases to construct a comprehensive biological network, thereby hindering the deciphering of key biological pathways and biomarkers for clinical translation. To address these limitations, we propose leveraging modern imaging technologies as an "intermediate bridge", because when critical biological pathways are triggered by genes, environmental factors, or their interactions, the earliest manifestations are impairments in cardiac and pulmonary structure and function (intermediate phenotypes). Accordingly, the DAILY project aims to enroll 50,000 participants across China, stratified by economic levels, geography, and living environments, to establish a high-quality bio-imaging database. This database will encompass: (1) advanced imaging-derived anatomical and functional phenotypes, along with precise hemodynamic measurements; (2) extensive multi-omics indicators, particularly genomics and downstream transcriptomics, proteomics, and metabolomics; (3) comprehensive living environments, psychological and cognitive date, and longitudinal health outcome; and (4) clinical medication and surgical records, along with other detailed clinical information.

Currently, there is a lack of a high-quality bio-imaging data platform based on the Chinese population to construct a complete pathway from genes/environment to disease, thereby enabling the development of promising strategies for CVD prevention and management.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Coronary CT angiography performed
* Informed consent acquired

Exclusion Criteria:

* Unable to complete the follow-up
* Serious chronic kidney disease (eGFR< 30 ml/min/1.73 m2)
* Serious liver disease or dysfunction (chronic active hepatitis and cirrhosis, or aspartate aminotransferase (AST) or alanine transaminase (ALT) > 3 times the upper limit of normal)
* Not appropriate to be tested due to birth planning, allergies, acute thyroid storm, etc.
* Suspected or known infectious diseases, such as hepatitis B virus (HBV), human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS), and Treponema pallidum (syphilis), etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutively enrolled individuals scheduled for coronary CTA, including those with known or suspected coronary artery disease (CAD) or individuals undergoing screening
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2038-05-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | Once a year until the tenth year
  Occurrence of major adverse cardiovascular events at prespecified follow-up ( once a year till the thirty year), defined as a composite of all-cause death, non-fatal myocardial infarction, unplanned revascularization , and hospitalization for unstable angina. Death cases consist of cardiovascular death, non-cardiovascular death, and undetermined cause of death.

SECONDARY OUTCOMES:
Invasive coronary angiography | Once a year until the tenth year
  Including invasive coronary angiography, diagnostic invasive coronary angiography with revascularization, and invasive coronary angiography without obstructive coronary disease (> 70% or >50% diameter stenosis)
Coronary revascularization | Once a year until the tenth year
  Coronary artery bypass grafting, percutaneous coronary interventions
Cardiovascular death, heart failure, atrial fibrillation, non-fatal MI, non-fatal stroke, unplanned revascularization, hospitalization for unstable angina | Once a year until the tenth year
  Cardiovascular death, heart failure, atrial fibrillation, non-fatal MI, non-fatal stroke, unplanned revascularization, hospitalization for unstable angina
Coronary plaque progression, regression, formation | Once every two years at least, until the tenth year
  Changes in the degree of coronary artery stenosis or plaque volume, or coronary plaque formation, or the volume, characteristics, and composition of high-risk plaques will be observed in participants with serial coronary CTA
Changes in functional small airways, pulmonary small vessels and emphysema volume | Once every two years at least, until the tenth year
  Patients undergoing serial chest CT scans were followed up to monitor changes in quantitative CT parameters, including emphysema volume, functional small airway volume, normal lung parenchyma volume and its percentage of total lung volume, as well as quantitative pulmonary small vessel metrics: the number of pulmonary vessels located at 6, 9, 12, 15, 18, 21, and 24 mm from the pleura across the entire lung, and the number of small vessels with a cross-sectional area less than 5 mm², or other relevant parameters
Emerging disease, regression or progression of established disease | Once a year until the tenth year
  Emerging diseases across various systems, such as metabolic disorders (e.g., hypertension, hyperlipidemia, hyperglycemia), cardiovascular diseases (e.g., hypertrophic cardiomyopathy, myocarditis), peripheral vascular diseases (e.g., deep vein thrombosis, arteritis), respiratory diseases (e.g., COPD, pulmonary hypertension), neurological disorders (e.g., dementia, Alzheimer's disease), malignancies (e.g., lung cancer, breast cancer), and diseases of other systems, will be documented. Additionally, the progression or regression of established disease will be recorded, for example, the development of diabetic retinopathy following the worsening of diabetes or the regression of impaired glucose tolerance, as well as the early surgical treatment of lung cancer or its recurrence in advanced stages.
Medication adjustment | Once a year until the tenth year
  Medication adjustment includes the increase or decrease of the drug dose and the new addition or discontinuation of medications after CCTA examination.
Medication regularly | once a year till the tenth year
  Taking medication regularly defined as the total number of days within the final month of a year during which established medication is taken (including Antiplatelet agents, Antihypertensive agents, Hypoglycemic agents, Lipid-lowering agents, Anti-inflammatory agents and and other agents).
Smoking, alcohol consumption, dietary habits, physical activity, symptoms, life quality | Once every five years until the tenth year
  A questionnaire-based follow-up that will mainly focus on smoking, alcohol consumption, dietary habits, physical activity, symptoms, and life quality (EQ-5D)
Anxiety and cognition | Once every five years until the tenth year
  A questionnaire-based follow-up that will mainly focus on anxiety and cognition
Adverse reactions to iodinated contrast agents | Within 1 hour and between 1 hour to 1 week after after contrast agent injection
  Acute adverse and late adverse reactions to iodinated contrast agents

CONTACTS AND LOCATIONS:
Overall Officials: Longjiang Zhang, MD, Principal Investigator — Jinling Hospital, Affiliated Hospital of Medical School, Nanjing University
Locations (1):
- Longjiang Zhang, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No